CLINICAL TRIAL: NCT03941743
Title: Prevention of Paclitaxel-Associated Neuropathy With Fingolimod: a Pilot Trial
Brief Title: Fingolimod in Preventing Paclitaxel-Associated Neuropathy in Patients With Breast Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: MC18C1; NCI-2019-02741 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); MC18C1 (Other: Mayo Clinic); P30CA015083 (NIH)
Record Dates: First submitted 2019-05-06; First posted 2019-05-08 (Actual); Last update posted 2023-07-21 (Actual); Status verified 2023-07

CONDITIONS: Breast Carcinoma
MeSH Terms: conditions — Breast Neoplasms | interventions — Fingolimod Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Prevention (fingolimod hydrochloride) (Experimental): Patients receive fingolimod hydrochloride PO QD starting the day before chemotherapy, the day of chemotherapy, and 1 day after chemotherapy for 12 weeks.
  Interventions: Drug: Fingolimod; Drug: Fingolimod Hydrochloride; Other: Questionnaire Administration

INTERVENTIONS:
Drug: Fingolimod — Given PO
Drug: Fingolimod Hydrochloride — Given PO
  Other Names: FTY-720; FTY720; Gilenya
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This trial phase I studies how well fingolimod works in preventing chemotherapy-induced nerve pain (neuropathy) in patients with breast cancer who are taking paclitaxel. Fingolimod acts by suppressing immune reactions in the brain. This study is being done to see if fingolimod can reduce neuropathy caused by paclitaxel.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To obtain preliminary data to support whether fingolimod hydrochloride (fingolimod) will prevent chemotherapy-induced peripheral neuropathy (CIPN) in patients receiving weekly adjuvant/neoadjuvant paclitaxel therapy.

SECONDARY OBJECTIVES:

I. To obtain pilot data regarding the possible relative toxicities related to fingolimod therapy in this study situation.

OUTLINE:

Patients receive fingolimod hydrochloride orally (PO) once daily (QD) starting the day before chemotherapy, the day of chemotherapy, and 1 day after chemotherapy for 12 weeks.

After the completion of study, patients are followed up at 6, 12, and 18 months.

ELIGIBILITY:
Inclusion Criteria:

* Ability to complete questionnaires by themselves or with assistance.
* Paclitaxel at a dose of 80 mg/m^2 given every week for a scheduled course of 12 weeks for treating breast cancer.
* Life expectancy >= 6 months.
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0, 1.
* Negative pregnancy test (serum or urine) done =< 14 days prior to registration, for persons of childbearing potential only.
* Provide written informed consent.

Exclusion Criteria:

* Previous exposure to paclitaxel (please note that it is acceptable for patients to receive non-neurotoxic chemotherapy, like doxorubicin hydrochloride (Adriamycin) and cyclophosphamide (AC), before or after the weekly paclitaxel and/or to receive concurrent anti-her 2 therapy).
* Any of the following because this study involves an agent that has known genotoxic, mutagenic and teratogenic effects:

  * Pregnant persons
  * Nursing persons
  * Persons of childbearing potential who are unwilling to employ adequate contraception.
* Previous diagnosis of diabetic or other peripheral neuropathy.
* Current or previous use of fingolimod.
* History of the following preexisting conditions: ischemic heart disease, cardiac arrest, cerebrovascular disease, uncontrolled hypertension, symptomatic bradycardia, macular edema, recurrent syncope, severe untreated sleep apnea, herpes simplex virus (HSV), varicella zoster virus (VZV), chronic hepatitis, tuberculosis, fungal infections, skin cancer, or diabetes.
* Myocardial infarction, unstable angina, stroke, transient ischemic attack (TIA), decompensated heart failure requiring hospitalization or class III/IV heart failure < 6 months prior to registration.
* History or presence of Mobitz type II second-degree or third-degree atrioventricular (AV) block or sick sinus syndrome, unless patient has a functioning pacemaker.
* History of a hypersensitivity reaction to fingolimod or any of the excipients including rash, urticarial, and angioedema upon treatment initiation.
* Baseline corrected QT (QTC) interval >= 450 ms (on electrocardiography [EKG]).
* Concurrent use of a class Ia or III antiarrhythmic.
* Drugs with a known risk of torsades de pointes.
* Concurrent use of beta blockers, calcium channel blockers or digoxin.
* Use of immunosuppressive, or immune-modulating therapies that may have immunosuppressive effects.
* Immunocompromised patients including patients known to be human immunodeficiency virus (HIV) positive.
* Uncontrolled intercurrent illness including, but not limited to:

  * Ongoing or active infection
  * Unstable angina pectoris
  * Cardiac arrhythmia
  * Or psychiatric illness/social situations that would limit compliance with study requirements.
* Receiving any other investigational agent.
* Family history of a genetic/familial neuropathy.
* Received a vaccine (inactivated) =< 14 days prior to registration.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2019-12-12 (Actual); Primary Completion 2020-06-05 (Actual); Study Completion 2021-11-23 (Actual)

PRIMARY OUTCOMES:
Serially measured total sensory neuropathy scores | Baseline up to 18 months
  Obtained from the 6 individual Quality of Life Questionnaire (QLQ)-Chemotherapy-Induced Peripheral Neuropathy (CIPN)20 questions that quantify numbness, tingling, and pain in the fingers (or hands) and toes (or feet). The hypothesis will be tested with the two-sided one sample t-test at a significance level of 10%. In the event that the distribution of the patient?s average total sensory neuropathy scores is not approximately normally distributed, then variable transformation or a nonparametric one-sample Wilcoxon signed-rank test will be considered as alternative approaches.

SECONDARY OUTCOMES:
Incidence of adverse events (AEs) | Up to 18 months
  Scored using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE), version (v) 5.0. Will be summarized by reporting the number and percentage of patients. The maximum grade for each type of AE will be recorded for each patient and data listings and frequency tables will be clinically reviewed to determine overall patterns, including AE attribution (possible, probable, and definite) to fingolimod. Additionally, the number and percentage of patients experiencing sensory neuropathy as defined by NCI CTCAE v5.0 will be tabulated by grade (none, mild, moderate, and severe); the proportion of patients experiencing >= grade 2 (moderate) CTCAE sensory neuropathy will estimated with the exact 90% confidence interval.

CONTACTS AND LOCATIONS:
Overall Officials: Charles L Loprinzi, Principal Investigator — Mayo Clinic
Locations (3):
- United States (3):
  - Mayo Clinic, Rochester, Minnesota
  - The Ohio State University, Columbus, Ohio
  - Virginia Commonwealth University/ Massey Cancer Center, Richmond, Virginia

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials.